CLINICAL TRIAL: NCT01447186
Title: Adaptation of the American Cancer Society (ACS) Early Detection of Prostate Cancer Patient Decision Aid for Spanish Speaking Men
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2011-0747; 11095006 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2011-10-03; First posted 2011-10-06 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer; Cancer
Keywords: Prostate cancer screening; Prostate Cancer; Patient Decision Aid; Spanish Speaking Men; Spanish-language slide set; Focus group; Interview; Survey
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Decision Aid for Spanish Speaking Men: Spanish-Language Slide Set
  Interventions: Behavioral: Post-Test Questionnaire; Behavioral: Interviews; Behavioral: Focus Groups

INTERVENTIONS:
Behavioral: Post-Test Questionnaire — Questionnaire following Demographic questionnaire, Pre-Test Knowledge Questionnaire and slide set review.
  Other Names: Surveys
Behavioral: Interviews — Using draft slide set, participants engage in think-aloud exercises, where each slide is reviewed and described.
Behavioral: Focus Groups — Up to 40 subjects will participate in the formative focus groups. Each group will be scheduled with 6 to 10 participants to explore Hispanic men's beliefs and concerns about prostate cancer and early detection.

SUMMARY:
Objectives:

The primary objective of this project is to develop and evaluate a Spanish-language slide set for administration in group settings, adapted from the content of the current guidelines and existing, self-administered ACS early detection decision aid.

A guide for educators will accompany the slide set so that materials may be distributed on a broad scale at the completion of the project. It is expected that these products will be made available to community-based educators and screening programs to be used in support of an IDM process for early detection of prostate cancer with Spanish-speaking men.

Specific Aims:

To conduct an extensive review of the literature and other resources to identify themes related to early detection, concerns and beliefs about prostate cancer in Hispanic men. Findings will be used to adapt the slideset.

To cognitive test the Spanish-language decision aid slide set with Hispanic men To conduct focus groups to evaluate the acceptability of the adapted slide set with Spanish-speaking Hispanic men who are candidates for prostate cancer screening. Participants will be tested for their knowledge of prostate cancer and acceptability of materials (e.g. length, clarity, amount and balance of information provided).

DETAILED DESCRIPTION:
Cognitive Testing Interviews:

If you agree to take part in this study, you will complete a questionnaire about your demographics (age, race, country of origin), education and family history of prostate cancer. This questionnaire should take about 5 minutes to complete.

Then you will take part in a one on one interview with a bilingual member of the study staff. You will be shown draft versions of a slide show about prostate cancer screening. You will then be asked to describe the information in the slides in your own words. You will also be asked about how easy or hard the information is to understand. The interview should last about 1 hour.

Length of Study:

Answering the questionnaire and participating in the interview will take about 1 to 1½ hours of your time. Your participation in this study will be over when the interview is complete.

Evaluation Focus Groups:

If you agree to take part in this study, you will complete 2 questionnaires about your demographics (age, race, country of origin), education, family history of prostate cancer, and knowledge of prostate cancer and its screening. These questionnaires should take about 10 minutes to complete. After the questionnaires, you will take part in a focus group with other men and members of the study.

In the focus group, a bilingual study staff member will lead the discussion by showing the group slides about prostate cancer screening. A doctor or healthcare professional designee will be available to answer questions about prostate cancer screening.

After viewing the slides, you will complete another questionnaire about what you know about prostate cancer. It will also ask what you thought about the information in the slides.

Length of Study:

Answering the questionnaires and participating in the focus group will take about 1 to 1½ hours of your time. Your participation in this study will be over when the focus group session is complete.

This is an investigational study.

Up to 60 participants will take part in this multicenter study. Up to 10 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male 45 years of age or older.
2. Ethnicity is Hispanic.
3. Language spoken is Spanish.

Exclusion Criteria:

1. Personal history of prostate cancer.
2. Active military personnel.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is Spanish-speaking Hispanic males, over 45 who have no personal history of prostate cancer who are or will soon be candidates for screening.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-09-21 (Actual); Primary Completion 2015-01-13 (Actual); Study Completion 2015-01-13 (Actual)

PRIMARY OUTCOMES:
Develop and Evaluate Spanish-Language Slide Set for Group Settings | At Completion of Focus Group, Questionnaire, and Interview - 1 1/2 hours
  For the evaluation aim of this study a Paired T-Test will be used before and after intervention measures of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org